CLINICAL TRIAL: NCT06282250
Title: An Explorative and Experimental Study to Assess the Feasibility, Acceptability, and Effectiveness of Early Intervention With Light, Lifestyle and ImCT Therapy in Individuals at Risk for Bipolar Disorder
Brief Title: Seeing the Light: Early Intervention in People at Risk for Bipolar Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geestelijke Gezondheidszorg Eindhoven (GGzE) (Other)
Responsible Party: Principal Investigator, Else Treffers, Principal investigator, Geestelijke Gezondheidszorg Eindhoven (GGzE)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: in progress
Record Dates: First submitted 2023-07-03; First posted 2024-02-28 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Bipolar Disorder; Mood Swing; Prodromal Symptoms
Keywords: Bipolar disorder; Early intervention; Light therapy; Early detection; Lifestyle; Imagery Focused Cognitive Therapy
MeSH Terms: conditions — Bipolar Disorder; Prodromal Symptoms | interventions — Ultraviolet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psycho-education and Imagery Focused Cognitive Therapy (in addition to Bright Light Therapy) (Other): Treatment will be personalized in accordance to one of three options:
  1. In case of depressive symptoms.
  Bright Light Therapy (BLT) will be administered for 30 minutes on five consecutive days (duration: 1-3 weeks).
  1 PE session focused on lifestyle and physical activity will take place. 6 sessions of ImCT will take place. This includes in-depth identification of images, constructing a micro-formulation along the lines of regular Cognitive Behavioural Therapy.
  2. In case of hyperactivity symptoms.
  The same PE and ImCT will be administered. The exception is that in this case, BLT is replaced by wearing blue-light blocking glasses for 1-3 weeks, 1 hour prior to bedtime.
  3. In case of at risk mental state, but no clear depressive or hyperactive symptoms.
  The same PE and ImCT will be administered. There will be no light intervention.
  Interventions: Behavioral: Bright light therapy + Psycho-education + Imagery focused Cognitive Therapy; Behavioral: Blue-light blocking glasses + Psycho-education + Imagery focused Cognitive Therapy; Behavioral: Psycho-education + Imagery focused Cognitive Therapy

INTERVENTIONS:
Behavioral: Bright light therapy + Psycho-education + Imagery focused Cognitive Therapy — Week 1-3: BLT will be administered for 30 minutes on five consecutive days, starting on Monday of the work week, between 7:30 AM and 10:00. The effect of the light therapy is evaluated by means of the Self-Rated Quick Inventory of Depressive Symptoms (QIDS-SR). Further treatment strategy is determined on the basis of these results:
  * If the patient has achieved remission (QIDS-SR < 6), BLT has been successful and the patient can continue with PE and IMCT.
  * If there is insufficient or no response (QIDS-SR of 6 or higher), BLT is extended with five more sessions the following week.
  * If necessary, a third week is optional.
  Week 2-4: Psycho Education will follow, 1 session.
  Week 3/4-9/10: ImCT will follow, 6 sessions.
Behavioral: Blue-light blocking glasses + Psycho-education + Imagery focused Cognitive Therapy — Week 1-3: blue-light blocking glasses will be administered. Week 2-4: Psycho Education will follow, 1 session.
  Week 3/4-9/10: ImCT will follow, 6 sessions.
Behavioral: Psycho-education + Imagery focused Cognitive Therapy — Week 1: Psycho Education, 1 session.
  Week 2-7: ImCT will follow, 6 sessions.

SUMMARY:
In the current study, the feasibility, acceptability and effectivity of a new add-on early intervention program for individuals at risk for the development of bipolar disorder is evaluated. This intervention program entails psycho-education, light and lifestyle therapy in combination with Imagery focused Cognitive Therapy (ImCT). The program aims to contribute to early intervention by focusing on subclinical mood swings, anxiety symptoms, circadian rhythm and lifestyle factors such as activity level. We hypothesize a relationship between this early intervention and a significant improvement in mood symptoms, anxiety, subjective and objective sleep factors and lifestyle variables. Also, the feasibility, acceptability and associations with clinical improvement of symptoms will be studied.

Additionally, in a separate validation study, data will be collected to validate a new instrument for the early detection of those at risk for bipolar disorders. The Semistructured Interview of At Risk Bipolar States (SIBARS) (Fusar-Poli et al., 2022) will be translated and validated in a Dutch sample, in cooperation with its creators, Prof. Dr. P. Fusar-Poli and colleagues.

DETAILED DESCRIPTION:
Severe mental illnesses (SMI) distinguished as bipolar disorder and psychotic spectrum disorders, substantially impair patients' engagement in functional and occupational activities and severely limit social and societal functioning (GGZ Standaarden, 2022; NIH, 2022; NIMH, 2018). Based on the Dutch definition of SMI 1.7% of the national population suffers from an SMI (GGZ Standaarden, 2022). Despite this, time between first symptoms and accurate SMI diagnosis, can add up to more than 9.5 years in the case of bipolar disorders. For the psychotic spectrum, an early detection and intervention program (UHR) carried out by special EDI-Teams already exists, and has been found effective in limiting the transition to SMI with fifty percent. For bipolar disorders, no such program exists. This raises the question whether prodromal and subclinical symptoms of this disorder can be detected earlier and if transition into SMI can be limited. In light of current studies into the at-risk mental state, and the current development towards a possible transdiagnostic model for early detection and intervention of SMI (CHARMS-categories; (Liu et al., 2022)), the current study aims to contribute to limiting the transition into bipolar disorder. As a disturbance in circadian rhythm, as well as mood and anxiety symptoms are risk indicators for SMI in general and bipolar in specific, the current study evaluates an early intervention program for individuals at risk for developing an SMI, with a focus on bipolar symptomatology.

Individuals at risk will answer questions from the SIBARS interview. As explained in a publication of Fusar-Poli et al. (2022), "The Semi-structured Interview for Bipolar At Risk States (SIBARS) included a combination of several items adapted from well-established rating scales: (CAARMS (Yung et al., 2005); Hypomania Checklist-32 (Angst et al., 2005); Altman Self-Rating Mania Scale (Altman et al., 1997); TEMPS-A questionnaire (Akiskal et al., 2005); QIDS-SR (Rush et al., 2003); Bergen Insomnia Scale (Pallesen et al., 2008); Idiopathic hypersomnia questionnaire (Vernet et al., 2010)). The SIBARS interview was developed for youths aged 15-35 and comprehended 5 domains: 1. Subtreshold Mania, 2. Depression, 3. Cyclothymic Features, 4. Genetic Risk, 5. Mood Swings. Subtreshold Mania, Depression and Mood Swings are continuous rating scales (that include a severity and frequency anchors), while Cyclothyimc Features and Genetic Risk are categorical scales (yes/no). The cut-offs allow assigning the specific subgroup of the BARS criteria: 1. Substreshold Mania, 2. Depression+Cyclothymic Features, 3. Depression+Genetic Risk, 4. Cyclothymic Features+Genetic Risk, 5.Subtreshold Mixed Episode, 6. Mood Swings."

ELIGIBILITY:
Inclusion Criteria:

* Must be bound to start the early intervention treatment being evaluated
* Aged 16-35, or > 35 by indication of the patients' treating clinician
* Found to be at risk for SMI, as determined by the Early Detection and Intervention Team of GGzE
* Sufficient knowledge of Dutch or English language
* Ability to give informed consent
* Willing to complete daily monitoring throughout the duration of the study

Exclusion Criteria:

* Learningdifficulties,organicbraindiseaseorsevereneurologicalimpairment.
* Previously received BLT (less than 3 weeks prior to study entry
* Current severe substance or alcohol misuse (clinicians' assessment)
* In case of BLT: eye problems contraindicating BLT and/or being unable to visit the GGzE

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptom scores on the IDS-SR | at baseline; 3 x per day during whole study (up to 7 weeks); immediately after intervention; and at 3 months follow-up
  Significant lowering of IDS-SR questionnaire scores
Change in hyperactive symptom scores on the ASRM | at baseline; 3 x per day during whole study (up to 7 weeks); immediately after intervention; and at 3 months follow-up
  Significant lowering of ASRM questionnaire scores
Change in anxiety symptom scores on the BAI | at baseline; 3 x per day during whole study (up to 7 weeks); immediately after intervention; and at 3 months follow-up
  Significant lowering of BAI questionnaire scores
Change in sleep quality subjective rating on 11-point Likert scale | at baseline; 3 x per day during whole study (up to 7 weeks); immediately after intervention; and at 3 months follow-up
  Significant improvement in subjective rating of sleep quality questionnaires
Change in activity levels subjective rating on 11-point Likert scale | at baseline; 3 x per day during whole study (up to 7 weeks); immediately after intervention; and at 3 months follow-up
  Changes in daily and pre-post intervention self-report measurement of activity levels

CONTACTS AND LOCATIONS:
Overall Officials: Inge Bongers, Prof. Dr., Principal Investigator — GGzE, Tilburg University
Locations (1):
- Geestelijke Gezondheidszorg Eindhoven (GGzE), Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The raw data is generated at the research location and is not shared with other researchers working elsewhere. After publication of the results, only data without privacy sensitive information and without study specific codes (fully anonymous), that support the findings are available from GGzE upon reasonable request (both in and outside the European Union). Before sharing this anonymous data, GGzE carefully investigates this request in consideration of the Dutch AVG and UAVG (Dutch Act on Implementation of the General Data Protection Regulation).
Supporting Information: Study Protocol
Time Frame: After pilot, June 2025, protocol will be expanded to multi-centre level.

REFERENCES:
- [Derived] Treffers E, Snaphaan L, van den Berg KC, Bongers IMB. A study protocol for the feasibility and acceptability of a personalized early intervention combining light therapy, lifestyle psychoeducation, and imagery-focused cognitive therapy in individuals at risk for bipolar disorder. Int J Bipolar Disord. 2026 Jan 22. doi: 10.1186/s40345-026-00410-4. Online ahead of print. PMID 41572055